CLINICAL TRIAL: NCT04476849
Title: A Phase 1 Open-label Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics, Safety and Tolerability of Fezolinetant Compared to Subjects With Normal Renal Function
Brief Title: A Study to Investigate the Effect of Renal Impairment on the Safety and Tolerability of Fezolinetant Compared to Participants With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2693-CL-0008
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers; Renal Impairment
Keywords: Healthy volunteers; Pharmacokinetics; ES259564; Renal impairment; fezolinetant
MeSH Terms: conditions — Renal Insufficiency | interventions — fezolinetant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Fezolinetant: Mild renal impairment (Experimental): Participants will receive a single oral dose of fezolinetant under fasting conditions on Day 1.
  Interventions: Drug: fezolinetant
- Fezolinetant: Moderate renal impairment (Experimental): Participants will receive a single oral dose of fezolinetant under fasting conditions on Day 1.
  Interventions: Drug: fezolinetant
- Fezolinetant: Severe renal impairment (Experimental): Participants will receive a single oral dose of fezolinetant under fasting conditions on Day 1.
  Interventions: Drug: fezolinetant
- Fezolinetant: Normal renal function (Experimental): Participants will receive a single oral dose of fezolinetant under fasting conditions on Day 1.
  Interventions: Drug: fezolinetant

INTERVENTIONS:
Drug: fezolinetant — Oral
  Other Names: ESN364

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of a single oral dose of fezolinetant and ES259564 (fezolinetant metabolite) in female participants with varying levels of renal impairment (mild, moderate and severe) compared to healthy female participants with normal renal function.

This study will also evaluate the safety and tolerability of a single oral dose of fezolinetant in female participants with varying levels of renal impairment (mild, moderate and severe) and healthy female participants with normal renal function.

Renal function will be measured by estimated glomerular filtration rate (eGFR) using the modification of diet in renal disease (MDRD) formula: Mild (eGFR 60 to < 90 mL/min per 1.73 m^2) renal impairment; moderate (eGFR 30 to < 60 mL/min per 1.73 m^2) renal impairment, severe (eGFR < 30 mL/min per 1.73 m^2) renal impairment and not on hemodialysis and normal (eGFR ≥ 90 mL/min per 1.73 m^2) renal function.

DETAILED DESCRIPTION:
This study will be comprised of four groups of participants based on renal function. Participants will be screened for up to 28 days prior to investigational product (IP) administration on Day 1. Eligible participants with mild, moderate and severe renal function and healthy participants with normal renal function will be admitted to the clinical unit on Day -1 and will be residential for a single period of six days/five nights. On Day 1, participants will receive a single oral dose of fezolinetant under fasting conditions followed by a 96-hour in-house blood and urine sampling period. Participants are to remain awake, seated or semirecumbent and avoid lying on either the left or right side for at least four hours postdose. Standard safety and tolerability assessments will be conducted. Participants will be discharged from the clinical unit on Day 5 on the condition that all required assessments have been performed and that there are no medical reasons for a longer stay in the clinical unit.

The study will be completed with an end-of-study visit (ESV). The ESV will take place five to nine days after the last pharmacokinetic sample is collected or at early discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Body Mass Index (BMI) range of 18.5 to 40 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Female subject is not pregnant and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance for at least 30 days prior to day -1 through at least 30 days after final IP administration
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
* Female subject must not donate ova starting from administration of IP and throughout the study period and for 30 days after final IP administration.
* Subject has normal renal function as defined by estimated glomerular filtration rate (eGFR) using the modification of diet in renal disease (MDRD) formula ≥ 90 milliliters per minute (mL/min) per 1.73 m^2 or subject has varying degrees of chronic kidney disease as defined by the National Kidney Foundation and by eGFR:

  * 60 to < 90 mL/min per 1.73 m^2 for subject with mild renal impairment
  * 30 to < 60 mL/min per 1.73 m^2 for subject with moderate renal impairment
  * < 30 mL/min per 1.73 m^2 and not on hemodialysis for subject with severe renal impairment
* Subject has adequate venous access.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has received any investigational therapy within 28 days or five half-lives, whichever is longer, prior to Day -1.
* Subject has any condition which makes the subject unsuitable for study participation.
* Female subject who has been pregnant within six months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to fezolinetant or any components of the formulation used.
* Subject has had previous exposure with fezolinetant.
* Subject has any of the liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST], and total bilirubin [TBL]) ≥ 1.5 × the Upper Limit of Normal (ULN) on Day -1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to IP administration.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to Day -1.
* Subject has smoked, used tobacco-containing products and nicotine or nicotine-containing products (e.g., electronic vapes) within six months prior to screening or the subject tests positive for cotinine at screening or on Day -1.
* Subject has a history of consuming > 7 units of alcoholic beverages per week within six months prior to screening or has a history of alcoholism three months prior to screening or drug/chemical/ substance abuse within one year prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol at screening or on Day -1.
* Subject has used any inducer of cytochrome P450 (CYP) 1A2 in the three months prior or inhibitors of CYP 1A2 in the two weeks or five half-lives, whichever is longer, prior to Day -1.
* Subject has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within seven days prior to Day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Subject has a positive serology test for hepatitis A virus antibodies (immunoglobulin M), hepatitis B core antibodies, hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Subject is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.

Additional criteria for subjects with renal impairment:

* Subject who has a history of any clinically significant illness (other than renal disease and conditions related to renal disease, such as stable diabetes and stable hypertension), medical condition or laboratory abnormality within 3 months prior to screening which precludes the subject from study participation.
* Subject has a mean pulse < 40 or > 90 beats per minutes (bpm); mean systolic blood pressure (SBP) < 90 or > 160 millimeters of mercury (mmHg); mean diastolic blood pressure (DBP) < 50 or > 100 mmHg (measurements taken in triplicate after subject has been resting in the supine position for at least five minutes; pulse will be measured automatically) on Day -1. If the mean blood pressure exceeds the limits above, one additional triplicate may be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) of > 480 msec on Day -1. If the mean QTcF exceeds the limits above, one additional triplicate ECG may be taken.
* Subject who has had a change in dose regimen of medically required medication(s) in the two weeks prior to IP administration (permitted concomitant medications) and/or subject for whom dose changes are likely to occur during the study (minor dose changes are allowed in agreement with the sponsor) and/or subject has used nonpermitted concomitant medication(s) (including vitamins, hormonal contraceptives, hormone replacement therapy [HRT] and natural and herbal remedies, e.g., St. John's Wort) in the three weeks prior to admission to the clinical unit.
* Subject who requires or is likely to require any new concomitant medications during the course of the study.
* Subject who has a renal disease secondary to malignancy.
* Subject who has a fluctuating or rapidly deteriorating renal function within four weeks prior to IP administration, as indicated by strongly varying or worsening clinical and/or laboratory signs of renal impairment within the screening period.
* Subject has a hemoglobin result of < 9 grams per deciliter.
* Subject has a functioning kidney transplant.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within three months prior to Day -1 or the subject tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) at screening or on Day -1, unless the positive result is due to an approved prescription medication.

Additional criteria for healthy subjects with normal renal function:

* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has any clinically significant abnormality following the physical examination, ECG and protocol-defined clinical laboratory tests at screening or on Day -1.
* Subject has a mean pulse < 45 or > 90 bpm; mean SBP > 150 mmHg; mean DBP > 90 mmHg (measurements taken in triplicate after subject has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on Day -1. If the mean blood pressure exceeds the limits above, one additional triplicate may be taken.
* Subject has a mean QTcF of > 450 msec on Day -1. If the mean QTcF exceeds the limits above, one additional triplicate ECG may be taken.
* Subject has used any prescribed or nonprescribed drugs (including vitamins, hormonal contraceptives, HRT and natural and herbal remedies, e.g., St. John's Wort) in the two weeks prior to IP administration, except for occasional use of acetaminophen (up to 2 g/day).
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within three months prior to Day -1 or the subject tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) at screening or on Day -1.
* Subject has creatinine level outside normal limits on Day -1. In such a case, the assessment may be repeated once.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of Fezolinetant in Plasma: Area Under the Concentration-time Curve (AUC) From the Time of Dosing Extrapolated to Time Infinity (AUCinf) | Up to 5 days
  AUCinf will be recorded from the PK plasma samples collected.
PK of Fezolinetant in Plasma: AUC From the Time of Dosing to the Last Measurable Concentration (AUClast) | Up to 5 days
  AUClast will be recorded from the PK plasma samples collected.
PK of Fezolinetant in Plasma: Maximum Concentration (Cmax) | Up to 5 days
  Cmax will be recorded from the PK plasma samples collected.
PK of Fezolinetant in Plasma: Apparent Clearance (CL/F) | Up to 5 days
  CL/F will be recorded from the PK plasma samples collected.
PK of Fezolinetant Metabolite ES259564 in Plasma: AUCinf | Up to 5 days
  AUCinf will be recorded from the PK plasma samples collected.
PK of Fezolinetant Metabolite ES259564 in Plasma: AUClast | Up to 5 days
  AUClast will be recorded from the PK plasma samples collected.
PK of Fezolinetant Metabolite ES259564 in Plasma: Cmax | Up to 5 days
  Cmax will be recorded from the PK plasma samples collected.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 14 days
  AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA). An AE is any untoward medical occurrence in a participant administered an IP and which does not necessarily have to have a causal relationship with this treatment.
Number of Participants With Laboratory Value Abnormalities and/or Adverse Events (AEs) | Up to 14 days
  Number of participants with potentially clinically significant laboratory values.
Number of Participants With Vital Sign Abnormalities and/or Adverse Events (AEs) | Up to 14 days
  Number of participants with potentially clinically significant vital sign values.
Number of Participants With 12-lead Electrocardiogram (ECG) Abnormalities and/or Adverse Events (AEs) | Up to 14 days
  Number of participants with potentially clinically significant 12-ECG values.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (7):
- United States (7):
  - National Institute of Clinical Research, Garden Grove, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism research, LLC, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.